CLINICAL TRIAL: NCT05609929
Title: A Phase I, Single-center, Open-label, Fixed Sequence Study in Chinese Healthy Male Adults to Evaluate the Effect of Omeprazole on the Pharmacokinetics of AB-106
Brief Title: Study the Effect of Omeprazole on AB-106 Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nuvation Bio Inc. (Industry)
Collaborators: AnHeart Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AB-106-C114
Record Dates: First submitted 2022-10-26; First posted 2022-11-08 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Pharmacokinetic Study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Omeprazole combined with AB-106 group (Experimental)
  Interventions: Drug: Multiple administration of omeprazole Single administration of AB-106

INTERVENTIONS:
Drug: Multiple administration of omeprazole Single administration of AB-106 — Take AB-106 capsule 400 mg orally on an empty stomach in the morning of the first day of the first cycle Take omeprazole magnesium enteric coated tablets 40mg once a day, 30 minutes before breakfast on days 1-4 of the second cycle. On the morning of the fifth day of the second cycle, the subjects will take omeprazole magnesium enteric coated tablets 40 mg, and AB-106 capsules 400 mg after an interval of 1 hour

SUMMARY:
This is a single-center, open-label, fixed sequence phase I clinical study. To evaluate the effect of continuous administration of omeprazole magnesium enteric coated tablets on PK after single dose AB-106 capsule administration in Chinese healthy male subjects. This study includes a screening period (1-28 days before administration), treatment period (34 days), and follow-up period ( after the last dose completed 7 ± 3 days). The treatment period of this study was divided into two periods, and the subjects were divided into two groups, 12 subjects in the first group and 10 subjects in the second group. The treatment method and research process of each group of subjects are the same. After the first group of subjects completes the second cycle and is evaluated by the investigator and sponsor, the second group of subjects can start administration. If there are no more than 4 subjects in the first group who have vomiting gastrointestinal reaction (vomiting occurs within 8 hours after each cycle of administration) after completing the two cycles of administration of AB-106 400 mg, they can be added to the second group of subjects, and the number of added subjects shall not exceed the number of subjects who have vomiting gastrointestinal reaction. If more than 4 subjects have gastrointestinal reaction of vomiting, the investigator and sponsor will make a comprehensive evaluation, and can reduce the dosage of AB-106 to 200 mg, and 22 subjects will be included in the trial at one time or supplemented in the second group to complete the 400 mg dose group

ELIGIBILITY:
Inclusion Criteria:

1. Chinese male healthy subjects (health refers to the state without clinically relevant abnormalities confirmed by medical history, physical examination, vital signs, 12 lead ECG and clinical laboratory examination).
2. The age at the time of signing the informed consent was between 18 and 55 years old (including the threshold).
3. When screening, the body weight was more than 50 kg, and the body mass index (BMI) was between 19 and 26 kg/m2 (including the cut-off value).
4. Subjects voluntarily signed the Informed Consent Form (ICF).
5. Subjects can communicate well with researchers and complete the study according to the protocol.
6. Male subjects with fertility agree that they and their sexual partners must take effective contraceptive measures during the study period and within 90 days after the last dose, and agree not to donate sperm during this period.

Exclusion Criteria:

1. Evidence or medical history (including drug allergy) of hematology, kidney, endocrine, lung, gastrointestinal, cardiovascular, liver, spirit, nerve or allergic diseases with clinical significance according to the judgment of the investigator.
2. According to the judgment of the researcher, abnormal laboratory tests with clinical significance (blood routine test, blood biochemical test [fasting], urine routine test, blood coagulation function test).
3. Systolic blood pressure<90 mmHg or ≥ 140 mmHg, diastolic blood pressure<50 mmHg or ≥ 90 mmHg, and the abnormality judged by the investigator is clinically significant.
4. People with eye diseases or people with a history of eye diseases who are considered by the investigator to increase the risk of the subject through eye examination.
5. 12 lead ECG showed QTcF>450 ms (msec) or QRS interval>120 msec.
6. Fever history within 5 days before administration.
7. People with positive detection of hepatitis B virus surface antigen (HBs Ag), hepatitis C virus antibody (HCV Ab), human immunodeficiency virus (HIV) antibody, or Treponema pallidum (TP) antibody.
8. The food or drug known to be used 28 days before screening is a powerful inhibitor of cytochrome P450 3A4 enzyme (CYP3A4); Known for use 28 days before screening Its drug is CYP3A4 potent inducer; The drug used 28 days before screening and during the study was CYP3A4 substrate with a narrow therapeutic window.
9. The food or drug known to be used 28 days before screening is the substrate of P-gp
10. Take Chinese herbal supplements within 28 days before screening; Take any clinical study drug within 3 months or 5 half lives (whichever is longer) before screening; Prescription drugs or over-the-counter drugs and dietary supplements were used within 14 days or 5 half lives (whichever is longer) before screening. As an exception, acetaminophen/paracetamol can be used in a dose of 1 g/day.
11. Those who have been vaccinated with live vaccine or attenuated vaccine within 28 days before the start of the trial.
12. Subjects were unwilling to stop the intake of caffeinated or purine containing foods (such as coffee, tea, cola, chocolate) in each administration cycle from 48 hours before the first administration to the end of the last PK sample collection.
13. The alcohol intake is more than 14 units/week (1 unit of alcohol is equivalent to 360 mL of beer, 150 mL of wine, or 45 mL of Baijiu), or the subject is unwilling to stop drinking alcohol in each administration cycle, from 48 hours before the first administration to the end of the last PK sample collection, or the alcohol breath test is positive.
14. Smoking ≥ 5 cigarettes a day, or the subject is unwilling/unable to stop nicotine intake in each dosing cycle from 48 hours before the first dosing to the end of the last PK sample collection.
15. Major surgery was performed within 6 months before administration.
16. Blood donation or blood loss ≥ 400 mL within 3 months before administration, or ≥ 200 mL within 1 month before administration
17. Suffer from gastrointestinal, liver, kidney diseases or other diseases or sequelae known to interfere with drug absorption, distribution, metabolism or excretion within 3 months before the screening period and during the screening period. A history of sensitivity to heparin or heparin induced thrombocytopenia.
18. Those who have a history of drug abuse or used soft drugs (such as marijuana) or hard drugs (such as heroin, cocaine, etc.) within one year before the study and during the study, or who are positive in drug screening.
19. Those who are unwilling or unable to comply with the lifestyle guidelines described in this program.
20. Staff of any institution affiliated to the clinical center and their immediate family members. Immediate relatives refer to those who are related by blood or law, including spouses, children, parents, brothers and sisters.
21. The researcher judged that it was not suitable to participate in the study

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Cmax | Day 1 to day15 for both treatment cycle one and cycle two, the total duration is 30 days
  plasma drug peak concentration
AUClast | Day 1 to day15 for both treatment cycle one and cycle two, the total duration is 30 days
  area under the plasma drug concentration time curve from 0 to the last measurable drug concentration time point
AUCinf | Day 1 to day15 for both treatment cycle one and cycle two, the total duration is 30 days
  Area under the plasma drug concentration time curve from 0 to infinity (if it can be calculated reliably)

SECONDARY OUTCOMES:
Tmax | Day 1 to day15 for both treatment cycle one and cycle two, the total duration is 30 days
  Time to reach plasma drug peak concentration
λ z | Day 1 to day15 for both treatment cycle one and cycle two, the total duration is 30 days
  Elimination rate constant
t1/2 | Day 1 to day15 for both treatment cycle one and cycle two, the total duration is 30 days
  elimination half-life
CL/F | Day 1 to day15 for both treatment cycle one and cycle two, the total duration is 30 days
  Apparent clearance
Vz/F | Day 1 to day15 for both treatment cycle one and cycle two, the total duration is 30 days
  apparent distribution volume
Number of adverse events as assessed by CTCAE 5.0 | Screening period (1-28 days before treatment), treatment period (34 days) and follow-up period (7 ± 3 days after the last visit). The total duration is about 69 days.
  Number of participants with treatment-related or not-related adverse events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided